CLINICAL TRIAL: NCT02551692
Title: Effects of Smoking Environments on Craving and Smoking
Brief Title: Effects of Smoking Environments on Craving and Smoking (CameraCue2.0)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00063505; 1R01DA038442 (NIH)
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Tobacco Use Cessation Devices; Nicotine; Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NRT (Placebo Comparator)
  Interventions: Drug: Nicotine Patch; Drug: Placebo Capsule
- VAR (Placebo Comparator)
  Interventions: Drug: Varenicline; Drug: Placebo Nicotine Patch
- PLAC (Placebo Comparator)
  Interventions: Drug: Nicotine Patch; Drug: Placebo Nicotine Patch; Drug: Placebo Capsule

INTERVENTIONS:
Drug: Nicotine Patch — Participants will wear 21mg/day patches for days 1-14. After day 14, participants will make a quit attempt continue to wear the 21mg/d patches for 6 weeks, then step down to 14mg/d patches for 2 weeks and finally step down 7mg/d for the last 2 weeks of treatment. Participants will also take a placebo capsule. During days 8-14, participants will undergo 2 cue-exposure sessions.
  Other Names: NicoDerm CQ
  Arms: NRT; PLAC
Drug: Varenicline — Varenicline (VAR) will be administered by titrating to steady state levels over a 7 day induction period (.5 mg once daily in Days 1-3; .5 mg twice daily on Days 4-7 and 1 mg twice daily on Days 8-14). Participants will continue on 1mg twice daily until the end of treatment (days 15-84). Participants will also wear a placebo patch. During days 8-14, participants will undergo 2 cue-exposure sessions.
  Other Names: Chantix
  Arms: VAR
Drug: Placebo Nicotine Patch — In the PLAC group, participants will receive placebo patches and placebo capsules for 14 days prior to quitting smoking. They will then switch to wearing a nicotine patch the morning of their quit day in order to provide them with the minimum standard of care. During days 8-14, participants will undergo 2 cue-exposure sessions.
  In the VAR group, participants will wear a placebo patch while taking varenicline.
  Arms: PLAC; VAR
Drug: Placebo Capsule — In the PLAC group, participants will receive placebo patches and placebo capsules for 14 days prior to quitting smoking. They will then switch to wearing a nicotine patch the morning of their quit day in order to provide them with the minimum standard of care. During days 8-14, participants will undergo 2 cue-exposure sessions.
  In the NRT group, participants will take a placebo capsule while wearing nicotine patches.
  Arms: NRT; PLAC

SUMMARY:
The goal of this study is to evaluate the effects of varenicline versus nicotine replacement versus placebo on personal smoking environment cue (PSE) reactivity. The results of this study will inform whether first-line pharmacotherapies for nicotine dependence (e.g. nicotine patch, varenicline) alter reactivity to environment cues. The investigators propose to identify 120 regular cigarette smokers who will complete 10 visits (1 screening visit, 1 training visit, 1 camera turn-in 2 cue exposure sessions and 4 post-quit medication check sessions). Smokers will be randomized to one of three medication conditions: placebo (PLAC; n=40), transdermal nicotine patch (NRT; n=40) or varenicline (VAR; n=40) in a double blind, double-dummy design. Reactivity variables (craving, latency to smoke, and smoke intake) will be entered into 3 (Medication: NRT, VAR, PLAC) x 2 (Environment: smoking, nonsmoking) repeated measures ANOVAs with random-effects. The investigators hypothesize that personal smoking, as compared to nonsmoking environments, will be associated with greater reactivity (i.e. increased craving and smoke intake; decreased latency to smoke). A Medication x Environment interaction will be characterized by decreased reactivity to smoking as compared to nonsmoking environments in the VAR and NRT groups as compared to the PLAC group.

ELIGIBILITY:
Inclusion criteria:

1. generally healthy [(i.e. ambulatory, not currently sick)]
2. between the ages of 18 and 60
3. smoking of at least 5 cig/day of a brand delivering ≥ 0.5 mg nicotine (FTC method) for > 1 year
4. an expired CO concentration of at least 10 ppm (to confirm inhalation) or urinary cotinine >1000 ng/mL (NicAlert = 6).
5. interest in quitting smoking within the timeframe of the experiment.
6. ability to identify 4 personal smoking and 4 personal non-smoking places.

Exclusion criteria:

1. immediate or no desire to quit smoking;
2. inability to attend all required experimental sessions;
3. use of psychoactive medications;
4. use of smokeless tobacco including e-cigarettes in the past 30 days;
5. current alcohol or drug abuse;
6. use of illegal drugs as measured by urine drug screen (excluding marijuana);
7. use of experimental (investigational) drugs;
8. current use of nicotine replacement therapy or other smoking cessation treatment;
9. Hypertension (systolic >140 mm Hg, diastolic >100 mm Hg, coupled with a history of hypertension); subjects with no previous diagnosis of hypertension may have a screening blood pressure up to 160/100. Participants with a history of hypertension may, however, be allowed to participate in the study if the study physician determines that the condition is stable, controlled by medication, and in no way jeopardizes the individual's safety;
10. Hypotension with symptoms (systolic <90 mm Hg, diastolic <60 mm Hg);
11. Coronary heart disease;
12. Lifetime history of heart attack;
13. Cardiac (heart) disorder (including but not limited to valvular heart disease, heart murmur, heart failure, arrhythmia); Abnormal EKG results suggestive of ischemia or undiagnosed cardiovascular disease please consider adding if it seems reasonable. For example, ST-segment depression or elevation, T-wave abnormalities, and lack of R wave are obtained with a 12-lead EKG).
14. Active skin disorder (e.g., psoriasis) within the last year, except minor skin conditions (including but not limited to facial acne, minor localized infections, and superficial minor wounds);
15. Medical condition that may contraindicate participation in the opinion of the investigator and study physician.(for example, EKG results)
16. Current psychiatric disease (with the exception of anxiety disorders, OCD and ADHD);
17. Suicidal ideation (within the past 10 years) or lifetime occurrence of attempted suicide;
18. Current depression - The Prime-MD will be used to screen for current (within 2 weeks) depression. Potential subjects who score >9 (or who score >0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") will be excluded from study participation, and, at the discretion of the study physician, referred to appropriate psychiatric treatment;
19. Bulimia or anorexia;
20. Significant adverse reaction to Chantix/Varenicline in the past;
21. Currently pregnant, breast feeding or likely to become pregnant;
22. History of seizure disorder.
23. A quit attempt within the last 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2016-01; Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McClernon, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 participants were withdrawn from the study prior to treatment assignment due to either loss of interest, lost to contact, or inability to complete baseline procedures per protocol.
Groups:
- Placebo (PLAC): Placebo Nicotine Patch: Participants will wear 21mg/day patches for days 1-14. After day 14, participants will make a quit attempt, continue to wear the 21mg patches for 6 weeks, then step down to 14mg patches for 2 weeks and finally step down 7mg/d for the last 2 weeks of treatment. Participants will also take a placebo capsule. During days 8-14, participants will undergo 2 cue-exposure sessions.
  In the PLAC group, participants will receive placebo patches and placebo capsules for 14 days prior to quitting smoking. They will then switch to wearing a nicotine patch the morning of their quit day in order to provide them with the minimum standard of care. During days 8-14, participants will undergo 2 cue-exposure sessions.
- Transdermal Nicotine Patch (NRT): Nicotine Patch: Participants will wear 21mg/day patches for days 1-14. After day 14, participants will make a quit attempt continue to wear the 21mg/d patches for 6 weeks, then step down to 14mg/d patches for 2 weeks and finally step down 7mg/d for the last 2 weeks of treatment. Participants will also take a placebo capsule. During days 8-14, participants will undergo 2 cue-exposure sessions.
  In the NRT group, participants will take a placebo capsule while wearing nicotine patches.
- Varenicline (VAR): Varenicline: Varenicline (VAR) will be administered by titrating to steady state levels over a 7 day induction period (.5 mg once daily in Days 1-3; .5 mg twice daily on Days 4-7 and 1 mg twice daily on Days 8-14). Participants will continue on 1mg twice daily until the end of treatment (days 15-84). Participants will also wear a placebo patch. During days 8-14, participants will undergo 2 cue-exposure sessions.
  In the VAR group, participants will wear a placebo patch while taking varenicline.
Period: Overall Study
Arm/Group | Placebo (PLAC) | Transdermal Nicotine Patch (NRT) | Varenicline (VAR)
Started | 31 | 27 | 30
Completed | 30 | 26 | 25
Not Completed | 1 | 1 | 5
Not completed — Lost to Follow-up | 0 | 1 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (PLAC) | Transdermal Nicotine Patch (NRT) | Varenicline (VAR) | Total
Number analyzed (Participants) | 31 | 27 | 30 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (11.6) | 47.4 (11.8) | 41.2 (11.9) | 44.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 15 | 44
  Male | 14 | 15 | 15 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 28 | 29
  Not Hispanic or Latino | 30 | 25 | 2 | 57
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 17 | 14 | 45
  White | 16 | 9 | 14 | 39
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 27 | 30 | 88

OUTCOME MEASURES:

1. Primary Outcome: Change in Craving Score During Cue Exposure Task
Description: Scores range from 0 (no craving) to 100 (extreme craving).
Time Frame: Cue Exposure 1 (beginning of week 3) to Cue Exposure 2 (end of week 3)
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo (PLAC) | Transdermal Nicotine Patch (NRT) | Varenicline (VAR)
Number analyzed (Participants) | 30 | 26 | 25
score on a scale | -11.17 (24.93) | -8.84 (28.3) | -14.29 (25.09)
Statistical Analysis 1: Comparison: Placebo (PLAC) vs Transdermal Nicotine Patch (NRT) vs Varenicline (VAR); Test type: Other; p = 0.534, ANOVA; Partial sum of squares = 855.65

2. Primary Outcome: Change in Latency to Smoke During Cue Exposure Task
Description: The latency is the interval between smoking one cigarette and wanting, craving, or needing another.
Time Frame: Cue Exposure 1 (beginning of week 3) to Cue Exposure 2 (end of week 3)
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo (PLAC) | Transdermal Nicotine Patch (NRT) | Varenicline (VAR)
Number analyzed (Participants) | 30 | 26 | 25
seconds | 30.22 (71.58) | 48.04 (95.79) | 65.15 (133.12)
Statistical Analysis 1: Comparison: Placebo (PLAC) vs Transdermal Nicotine Patch (NRT) vs Varenicline (VAR); Test type: Other; p = 0.26, ANOVA; Partial sum of squares = 29602.69

3. Primary Outcome: Change in Smoke Intake During Cue Exposure Task
Description: Measured by number of puffs.
Time Frame: Cue Exposure 1 (beginning of week 3) to Cue Exposure 2 (end of week 3)
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: puffs
Arm/Group | Placebo (PLAC) | Transdermal Nicotine Patch (NRT) | Varenicline (VAR)
Number analyzed (Participants) | 30 | 26 | 25
puffs | 14.42 (6.35) | 12.21 (4.42) | 12.98 (7.90)
Statistical Analysis 1: Comparison: Placebo (PLAC) vs Transdermal Nicotine Patch (NRT) vs Varenicline (VAR); Test type: Other; p = 0.318, ANCOVA; Partial sum of squares = 101.69

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Placebo (PLAC) | Transdermal Nicotine Patch (NRT) | Varenicline (VAR)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/27 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/31 | 0/27 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/27 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PLAC) (N=31) | Transdermal Nicotine Patch (NRT) (N=27) | Varenicline (VAR) (N=30)
Bacterial blood infection (Infections and infestations) | 1 | 0 | 0
Blood in urine (Renal and urinary disorders) | 1 | 0 | 0
Dehydration (General disorders) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT02551692/Prot_SAP_000.pdf